CLINICAL TRIAL: NCT00270049
Title: The Effect of Subcutaneous r-HuEPO in Patients With Chronic Lymphocytic Leukemia
Brief Title: Epoetin Alfa for the Treatment of Anemia Resulting From Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005905
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-01

CONDITIONS: Anemia; Leukemia, Lymphocytic, Chronic; Leukemia, Lymphocytic; Cancer; Neoplasms; Quality of Life
Keywords: Anemia; cancer; leukemia; chronic lymphocytic leukemia; lymphocytic leukemia; epoetin alfa; erythropoietin; red blood cells; transfusions; quality of life
MeSH Terms: conditions — Anemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid; Neoplasms; Leukemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effect of treatment with epoetin alfa versus placebo on the percentage of red blood cells in anemic patients with chronic lymphocytic (white blood cell) leukemia and its effect on the patients' quality-of-life. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy, or both. Quality of life is also affected, in part because of the fatigue associated with anemia. Previous studies with epoetin alfa have suggested that achieving a higher hemoglobin level may improve the quality of life and help patients live longer. This is a 12-week, double-blind, placebo-controlled, multicenter study to determine the effect of treatment with epoetin alfa on the percentage of red blood cells in anemic patients with chronic white blood cell leukemia. At the start of the study, patients were either receiving no chemotherapy, single-agent chemotherapy, and/or were on prednisone (steroid) treatment. Patients will be randomly assigned 2:1 to receive either epoetin alfa or placebo. Patients receiving epoetin alfa will receive subcutaneous (under the skin) epoetin alfa injections 3 times per week and patients on placebo will receive an equal volume of matching placebo, injected subcutaneously 3 times per week. Based on patients' rate of increase in red blood cell percentage, the original dose of 150 units per kilogram 3 times per week may be raised gradually to 300 units per kilogram 3 times per week, to reach a target red blood cell percentage of 38% to 40%. Patients achieving the target red blood cell percentage will be eligible for a 12-week open-label extension of the study, which will focus on safety findings. Effectiveness will be determined by the proportion of patients who reach the target red blood cell percentage of 38% to 40% by the end of the study, the number of transfusions required, the proportion of patients achieving a red blood cell percentage of 38% to 40% at any time during the study, and changes in quality of life parameters. Safety evaluations, including the incidence of adverse events, laboratory tests, and vital signs, will be performed throughout the study. The hypothesis of the study is that epoetin alfa will be superior to placebo in increasing the percentage of red blood cells to the target level, reducing the number of transfusions required, and improving the quality of life. Epoetin alfa 150 units per kilogram 3 times weekly subcutaneously for 12 weeks. Individualized dose increases of 50 mg/week depend on red blood cell response, up to a maximum 300 units per kilogram 3 times per week to obtain the target level of 38% to 40% red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lymphocytic (white blood cell) leukemia
* having received either no cancer treatment, or treated with single-agent chemotherapy and/or prednisone for one month or a combination chemotherapy regimen
* having a Performance score of 0 (fully active, no disease restriction) to 3 (capable of only limited self-care, confined to bed or chair more than 50% of waking hours)
* having a life expectancy of at least 6 months
* having a hematocrit of <32%, a corrected reticulocyte count of <3%, platelets >25,000 cells/millimeter cubed, creatinine <2.0 mg/mL, a negative Coombs test (test for antibodies to red blood cells) and no occult blood in the stool

Exclusion Criteria:

* Patients with a clinically significant disease besides cancer
* having uncontrolled high blood pressure or a history of seizures
* received androgen therapy within 2 months of study
* received a transfusion within 1 week of study entry
* received radiation therapy within 1 month of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 1990-11; Study Completion 1994-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who reach the target of 38% to 40% red blood cells at the end of the study; Safety including the incidence of adverse events

SECONDARY OUTCOMES:
Transfusion requirements; Proportion of patients achieving red blood cell percentage of 38% to 40% any time during the study (unrelated to transfusions); Quality of life (physician's global assessment and patient's ability to perform daily activities)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Epoetin Alfa for Anemia From Chronic Lymphocytic Leukemia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=681&filename=CR005905_CSR.pdf